CLINICAL TRIAL: NCT00904397
Title: A Randomized, Open-Label Study Comparing the Efficacy and Safety of Lidocaine Patch 5% With Celecoxib 200 mg in Patients With Chronic Axial Low Back Pain
Brief Title: Lidocaine Patch 5% Versus Celecoxib 200 mg in Chronic Axial Low Back Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Rofecoxib was withdrawn from the market due to safety concerns.
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3220-013
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Lidoderm; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Lidoderm (Experimental): Lidocaine patch 5% (Lidoderm®, Endo Pharmaceuticals Inc.), 2 patches applied once daily (q24h) directly to the most painful area of the low back
  Interventions: Drug: Lidoderm®
- Celecoxib (Active Comparator): Celecoxib (Celebrex®, G.D. Searle & Co., Chicago, IL), one 200 mg oral capsule QD
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Lidoderm® — Patients participated in a 14-day washout period followed by a 12-week active treatment period. Eligible patients were randomized equally to one of two groups: lidocaine patch 5% or celecoxib 200 mg.
  Other Names: Lidocaine patch 5%
  Arms: Lidoderm
Drug: Celecoxib — Patients participated in a 14-day washout period followed by a 12-week active treatment period. Eligible patients were randomized equally to one of two groups: lidocaine patch 5% or celecoxib 200 mg.
  Arms: Celecoxib

SUMMARY:
Patients who had axial lower back pain (LBP) with or without radiation present for at least 3 months and had daily moderate to severe LBP as the primary source of pain participated in a Phase IV clinical trial to assess the efficacy of lidocaine patch 5% compared to celecoxib 200 mg in treating chronic axial LBP with and without radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Had axial LBP with or without radiation present for at least 3 months as defined below:

   * Chronic axial LBP without radiation: pain isolated to the axial low back without radiation into the buttock or below
   * Chronic axial LBP with radiation: pain that radiated to the buttock or below. This patient group could include patients with radicular/neuropathic and non-radicular components with leg pain component <50%
2. Had daily moderate to severe LBP as the primary source of pain
3. Had a normal neurological examination, including:

   * Motor strength
   * Sensory exam in lower extremities
   * Deep tendon reflexes
4. Had a normal 12-lead electrocardiogram (ECG) without any clinically significant abnormalities in heart rate, rhythm, or conduction
5. Had discontinued use of all analgesic medications (including over-the-counter [OTC] analgesics), glucosamine, and chondroitin prior to randomization (patients were allowed limited use of analgesic medications for indications other than non-study pain
6. At the baseline visit, patients were randomized to active treatment if they had an average daily pain intensity score of 5 or greater (on a 0 to 10 scale) for at least 3 days out of the 5 consecutive days immediately prior to the baseline visit; 0 was defined as "no pain" and 10 was defined as "pain as bad as ever imagined" as measured by Question 5 of the Brief Pain Inventory (BPI) and recorded in a diary

Exclusion Criteria:

1. Had spinal stenosis with >50% leg pain component
2. Had any other chronic pain condition that, in the opinion of the investigator, would interfere with patient assessment of LBP relief
3. Had a history of one or more back surgeries within 1 year of study entry
4. Had a moderate or greater hepatic impairment
5. Had a severe renal insufficiency (creatinine clearance of <30 mL/min)
6. Had experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs)
7. Had a prior history of peptic ulcer disease and/or gastrointestinal (GI) bleeding
8. Were taking analgesic medications that could not be discontinued during the study. Patients taking these medications prior to the study were required to discontinue use for the duration of the study. Patients using opioid analgesics at study entry were required to taper off these medications.
9. Were taking long-acting opioids or opioids that could not be discontinued over the first 5 days of the washout period
10. Were receiving fluconazole or lithium (secondary to drug-drug-interaction risks with celecoxib)
11. Had received an epidural steroid/local anesthetic injection within 4 weeks prior to study entry
12. Had received trigger point injections within 2 weeks prior to study entry
13. Had received Botulinum Toxin (Botox) injections for LBP within 6 months prior to study entry
14. Were using a lidocaine-containing product that cannot be discontinued during the study
15. Were using any topical medication applied to the low back region
16. Had previously failed treatment with Lidoderm analgesic patch for LBP
17. Had previously failed treatment with celecoxib or with any two COX-2 specific inhibitors other than celecoxib
18. Were taking class I anti-arrhythmic (e.g. mexiletine, tocainide)
19. Had a history of alcohol or substance abuse within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-07; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Week 12 in BPI average pain intensity score (Question 5). | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)

SECONDARY OUTCOMES:
Mean change from baseline to Weeks 2, 4, 6, 8, and 12 in daily pain intensity score as measured by Questions 3, 4, 5, and 6 of the BPI | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Mean change from baseline to Weeks 2, 4, 6, 8, and 12 in BPI pain relief score (Question 8). | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Mean change from baseline to Weeks 2, 4, 6, 8, and 12 in PQAS composite scores | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Mean change from baseline to Weeks 2, 4, 6, 8, and 12 in Oswestry Disability Index composite scores | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Investigator's Global Impression of Change in LBP at Week 12 (or premature discontinuation) | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Patient's Global Impression of Change in LBP at Week 12 (or premature discontinuation) | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Investigator's Global Assessment of Treatment Satisfaction at Week 12 (or premature discontinuation) | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Patient's Global Assessment of Treatment Satisfaction at Week 12 (or premature discontinuation) | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Safety assessments included AEs (including discontinuation due to AEs). | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Safety assessments included dermal assessment (lidocaine group only), skin sensory testing (lidocaine group only), clinical laboratory test results (including urinalysis, vital signs measurements, physical and neurological examinations, and body weight. | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)
Safety assessments included plasma lidocaine concentrations (lidocaine group only). | Visit - V2 (Day 0), V3 (Day 14), V4 (Day 28), V5 (Day 42), V6 (Day 56), V7 (Day 84)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Study Director — Endo Pharmaceuticals
Locations (21):
- United States (21):
  - Northport, Alabama
  - Phoenix, Arizona
  - Beverly Hills, California
  - Encinitas, California
  - San Diego, California
  - Spring Valley, California
  - Longwood, Florida
  - North Miami Beach, Florida
  - Plantation, Florida
  - Chicago, Illinois
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Berlin, New Jersey
  - Bethpage, New York
  - Tonawanda, New York
  - Charlotte, North Carolina
  - Dayton, Ohio
  - Allentown, Pennsylvania
  - Sellersville, Pennsylvania
  - Greer, South Carolina
  - Spokane, Washington